CLINICAL TRIAL: NCT01151982
Title: Primary Prevention of Major Depression Based on the Level and Profile of Risk of Primary Care Attenders: Cluster, Controlled, Randomised Trial
Acronym: predictD-CCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Carlos III Health Institute (Other Government); Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Juan Ángel Bellón Saameño, PhD Medicine, The Mediterranean Institute for the Advance of Biotechnology and Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PS09/00081
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Depression
Keywords: Depression; Primary prevention.; Primary health care.; Randomised controlled trial.
MeSH Terms: conditions — Depression | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial Intervention (Experimental): The intervention we propose to test has 3 actives components. The first one is the fact of giving information to the GPs about the level and risk profile of depression of their patients. The second one is the transmission of this information from the GP to the patient. The third one is the interaction GP/Patient once both have the information about the risk profile of depression and the psychoeducational intervention that the GP will provide to the patient.
  We will develop psychoeducational booklet, DVDs and websites for patients included in the intervention group.
  The psychoeducative intervention will be tailored to each patient based on his/her profile, risk level and patients' risk factors.
  The GPs will receive a 20-hours training course in the intervention. Moreover, we will assume a communitarian view, considering the patient as an active agent for change (empowerment). That is, GPs and patients will work together in order to promote patients' resources.
  Interventions: Behavioral: Psychosocial Intervention
- Usual Care (No Intervention): The kind of care that general practitioners usually provide when not knowing the level and risk profile of depression of the patients

INTERVENTIONS:
Behavioral: Psychosocial Intervention — The intervention we propose to test has 3 actives components. The first one is the fact of giving information to the GPs about the level and risk profile of depression of their patients. The second one is the transmission of this information from the GP to the patient. The third one is the interaction GP/Patient once both have the information about the risk profile of depression and the psychoeducational intervention that the GP will provide to the patient.
  We will develop psychoeducational booklet, DVDs and websites for patients included in the intervention group.
  The psychoeducative intervention will be tailored to each patient based on his/her profile, risk level and patients' risk factors.
  The GPs will receive a 20-hours training course in the intervention. Moreover, we will assume a communitarian view, considering the patient as an active agent for change (empowerment). That is, GPs and patients will work together in order to promote patients' resources.
  Arms: Psychosocial Intervention

SUMMARY:
The main objective is to measure the effectiveness of a new intervention for primary prevention of major depression based on the level and profile of risk of primary care attendees. Among the secondary objectives is to evaluate the cost-effectiveness and cost-utility of the intervention versus usual care. METHODS: This is a cluster, randomised controlled trial of a community intervention with cluster at the level of practice. It will be undertaken in primary medical care in 7 Spanish cities and 5 autonomous communities.The aim is to evaluate a new intervention for primary prevention of major depression based on patients' level and profile of risk. Family doctors in the intervention practices will provide the intervention for patients at risk. Patients at risk who are recruited in control practices will receive usual primary care. The main outcome is the accumulated incidence of major depression (measured by CIDI) during the follow-up. The investigators will assess main outcomes and other covariables at baseline, 6, 12, and 18 months. A random sample of 3,381 primary care attendees (1,690 for each arm), aged 18-75 and without major depression will be recruited in 70 health centres (140 family doctors) in 7 cities. The investigators shall undertake a logistic regression multilevel model with 4 levels (time, patient, doctor and health centre). The investigators shall also undertake multivariate gamma and quantile regression to assess respectively the cost-effectiveness and cost-utility of the new intervention versus usual care, estimating their standard errors by bootstrap.

ELIGIBILITY:
Inclusion Criteria:

* Patients among those attending to primary care centers.

Exclusion Criteria:

* Age under 18 or over 75 years.
* Unable to understand or speak Spanish.
* Represented patients (that is, someone else comes to visit on behalf of the patient).
* Cognitive impairment.
* Psychosis.
* Terminal illness.
* Planning to be outside of the the city during 4 or more months during the next 18 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3326 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Accumulated incidence of major depression | 18 months

SECONDARY OUTCOMES:
Cost-effectiveness and cost-utility | 18 months
  To evaluate the cost-effectiveness and cost-utility of the intervention versus usual care.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Servicio Andaluz de Salud. Distrito Sanitario Málaga, Málaga, Málaga
  - Málaga, Málaga

REFERENCES:
- [Derived] Fernandez A, Mendive JM, Conejo-Ceron S, Moreno-Peral P, King M, Nazareth I, Martin-Perez C, Fernandez-Alonso C, Rodriguez-Bayon A, Aiarzaguena JM, Monton-Franco C, Serrano-Blanco A, Ibanez-Casas I, Rodriguez-Sanchez E, Salvador-Carulla L, Garay PB, Ballesta-Rodriguez MI, LaFuente P, Del Mar Munoz-Garcia M, Minguez-Gonzalo P, Araujo L, Palao D, Gomez MC, Zubiaga F, Navas-Campana D, Aranda-Regules JM, Rodriguez-Morejon A, de Dios Luna J, Bellon JA. A personalized intervention to prevent depression in primary care: cost-effectiveness study nested into a clustered randomized trial. BMC Med. 2018 Feb 23;16(1):28. doi: 10.1186/s12916-018-1005-y. PMID 29471877
- [Derived] Bellon JA, Conejo-Ceron S, Moreno-Peral P, King M, Nazareth I, Martin-Perez C, Fernandez-Alonso C, Rodriguez-Bayon A, Fernandez A, Aiarzaguena JM, Monton-Franco C, Ibanez-Casas I, Rodriguez-Sanchez E, Ballesta-Rodriguez MI, Serrano-Blanco A, Gomez MC, LaFuente P, Munoz-Garcia Mdel M, Minguez-Gonzalo P, Araujo L, Palao D, Bully P, Zubiaga F, Navas-Campana D, Mendive J, Aranda-Regules JM, Rodriguez-Morejon A, Salvador-Carulla L, de Dios Luna J. Intervention to Prevent Major Depression in Primary Care: A Cluster Randomized Trial. Ann Intern Med. 2016 May 17;164(10):656-65. doi: 10.7326/M14-2653. Epub 2016 Mar 29. PMID 27019334
- [Derived] Bellon JA, Conejo-Ceron S, Moreno-Peral P, King M, Nazareth I, Martin-Perez C, Fernandez-Alonso C, Ballesta-Rodriguez MI, Fernandez A, Aiarzaguena JM, Monton-Franco C, Ibanez-Casas I, Rodriguez-Sanchez E, Rodriguez-Bayon A, Serrano-Blanco A, Gomez MC, LaFuente P, Del Mar Munoz-Garcia M, Minguez-Gonzalo P, Araujo L, Palao D, Espinosa-Cifuentes M, Zubiaga F, Navas-Campana D, Mendive J, Aranda-Regules JM, Rodriguez-Morejon A, Salvador-Carulla L, de Dios Luna J. Preventing the onset of major depression based on the level and profile of risk of primary care attendees: protocol of a cluster randomised trial (the predictD-CCRT study). BMC Psychiatry. 2013 Jun 19;13:171. doi: 10.1186/1471-244X-13-171. PMID 23782553